CLINICAL TRIAL: NCT06211192
Title: Evaluation of the Determinant Factors of Ceasing Anti-seizure Medication in Infants With Neonatal Seizures: A Single-center Retrospective Study
Brief Title: What Are the Determinant Factors of Ceasing Anti-seizure Medication in Infants With Neonatal Seizures?
Status: Completed | Type: Observational
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, İpek Dokurel, Medical Doctor, Balikesir University
Other Study IDs: YDKtreat
Record Dates: First submitted 2023-12-19; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Neonatal Seizure
Keywords: Neonate; Seizure; Early onset epilepsy; anti-seizure medication; acute provoke seizure
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: the first group consisted of infants who continued to receive ASM treatment after 12 months of age (referred to as "infants still on ASM after 12 months", n=69)
  Interventions: Other: retrospective data collection
- Group 2: the second group consisted of infants who had stopped ASM treatment before 12 months of age (referred to as "infants who had ceased ASM before 12 months", n=88)
  Interventions: Other: retrospective data collection

INTERVENTIONS:
Other: retrospective data collection — retrospective data collecting from medical records

SUMMARY:
The investigators aimed to determine the factors for ceasing anti-seizure medication in infants who experienced seizures during the neonatal period. This retrospective, single-center, descriptive study was conducted in Balıkesir between December 2020 and February 2023, and 157 neonates were recruited.

DETAILED DESCRIPTION:
This retrospective, single-center, descriptive study was conducted at the Department of Paediatric Neurology between December 2020 and February 2023, and 157 neonates were recruited to determine the factors related to ceasing ASM treatment in infants at a follow-up 2 years. According to the International League Against Epilepsy (ILAE) classification of neonatal seizures and their etiology, patients who were diagnosed with such seizures and received anti-seizure medication within the first 28 days of life were followed until their ASM was ceased after they were discharged from the neonatal intensive care unit. Infants are defined as children aged younger than 12 months. During this stage of neuronal development, the central nervous system is more susceptible to the harmful effects of external factors. Consequently, the investigators have planned to evaluate the study's initial 12-month follow-up results for our group. Afterwards, the infants were divided into two groups: the first group consisted of infants who continued to receive ASM treatment after 12 months of age (referred to as "infants still on ASM after 12 months", n=69); the second group consisted of infants who had stopped ASM treatment before 12 months of age (referred to as "infants who had ceased ASM before 12 months", n=88).

ELIGIBILITY:
Inclusion Criteria:

* Neonates with seizures diagnosed clinically or with conventional electroencephalography (cEEG) confirmation were enrolled.

Exclusion Criteria:

* with abnormal paroxysmal events that weren't determined to be seizures by cEEG, amplitude integrated EEG (aEEG) and video records,
* stopped medications due to their parents' decisions,
* with missing hospital records,
* delivered from pregnancies by assisted reproductive techniques were not enrolled.

Ages: 1 Hour to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants are defined as children aged younger than 12 months.According to the International League Against Epilepsy (ILAE) classification of neonatal seizures and their aetiology, patients who were diagnosed with such seizures and received anti-seizure medication within the first 28 days of life were followed until their ASM was ceased after they were discharged from the neonatal intensive care unit.
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
compile risk elements linked to extended use of anti-seizure medication retrospectively | 1-2 years
  Collecting the risk elements associated with long-term usage of anti-seizure medication from the participants' medical records in a retrospective manner.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Kösecik, Prof, Study Chair — Balikesir Üniversite Medical faculty hospital
Locations (1):
- Orkun Çetin, Balıkesir, Altieylul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided